CLINICAL TRIAL: NCT05377151
Title: A Dietitian-led Cluster Randomised Controlled Trial on the Effectiveness of mHealth Education on Health Outcomes Among Pregnant Women
Brief Title: Effectiveness of mHealth Education on Health Outcomes Among Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Chan Yoke Mun, Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 03210224
Record Dates: First submitted 2022-04-24; First posted 2022-05-17 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Pregnant Women
Keywords: Pregnant mother; Mobile health (mHealth); Nutrition and diet; Gestational Weight Gain; Quality of Life; Pregnancy outcomes
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mobile application (mHealth) intervention only (Experimental): - the subjects will receive mobile application (mHealth) intervention only
  Interventions: Other: Mobile application
- mobile application (mHealth) intervention and dietitian consultation (Experimental): - the subjects will receive the information from both mobile application (mHealth) and dietitian consultation
  Interventions: Other: Mobile application
- standard usual care- dietitian consultation (No Intervention): - the subjects will receive all the related information from the standard usual care- dietitian consultation

INTERVENTIONS:
Other: Mobile application — Nutrition intervention using either mHealth interventions or conventional methods will be carried out among pregnant women).
  Subjects will be allocated into three groups, namely, two interventions group which are:
  Group 1: mHealth intervention group (98 subjects)
  Group 2: mHealth intervention group + dietitian consultation (98 subjects)
  Group 3: control group (98 subjects)
  Arms: mobile application (mHealth) intervention and dietitian consultation; mobile application (mHealth) intervention only

SUMMARY:
Gestational weight gain (GWG), weight gain of a mother during pregnancy, is an important determinant that influence the health outcomes of mothers and fetus. There is an increasing trend of pregnant women using mobile health (mHealth) to assess for pregnancy-related health information. While evidence on the effectiveness of mHealth education on improving pregnancy outcomes among pregnant women is growing, the findings had been inconclusive with scarcity of such data in Malaysia. The objective of the study is to determine the effectiveness of a 9-month mHealth intervention on GWG and other outcomes (prenatal knowledge, physical activity, psychosocial well-being, nutritional status, quality of life and sleep quality) among pregnant women.

DETAILED DESCRIPTION:
This study will evaluate the usability, feasibility and practicality of a previously developed smartphone application with complete alpha and beta testing on pregnancy outcomes in a cluster randomised control trial (RCT).

The study will be completed by involving the nutrition intervention using either mHealth interventions or conventional methods that will be carried out among pregnancy women.

Subjects will be allocated into groups according to respective health clinics, namely, two interventions group which are:

Group 1: mHealth intervention group

Group 2: mHealth intervention group + dietitian consultation

Group 3: control group

which total of 294 eligible subjects will be recruited, with 98 subjects are needed in respective groups.

This is a cluster-randomised controlled trial. For Malaysia consist of two regions which are East Malaysia and West (or peninsular) Malaysia and they are actually about 400 miles (640 km) apart. At East Malaysia, we targeted on the area with higher density of population which are Klang Valley (Kuala Lumpur, Selangor and Putrajaya). As shown in Figure 1, for three states under Klang Valley, we obtained ethics approval from the Jabatan Kesihatan Negeri Selangor for Selangor state and Jabatan Kesihatan Wilayah Persekutuan Kuala Lumpur dan Putrajaya for Putrajaya state. In order to prevent cross contamination between the states, we use simple random sampling which Selangor been allocated into control group and Putrajaya as intervention group.

As under Putrajaya states only two clinics granted approval for data collection which are Presint 9 Health Clinic and Presint 18 Health Clinic. By using cluster sampling method, Presint 9 Health Clinic was randomised into intervention group 1 which whole cluster participant will be receiving mHealth intervention alone and Presint 18 Health Clinic into intervention group 2 which whole cluster participants will receive mHealth intervention group in addition with personal dietitian consultation.

There are nine districts in Selangor: Gombak, Hulu Langat, Hulu Selangor, Klang, Kuala Langat, Kuala Selangor, Petaling, Sabak Bernam and Sepang which consist of total of 81 health clinics, we stratified the number of health clinics within the 25 km radius from the Faculty of Medicine and Health Sciences, Universiti Putra Malaysia due to the geographical proximity and financial constraints (limited budget). There were total of 15 health clinics after stratification and simple random sampling was done which Seri Kembangan health clinics in Petaling District had been chosen as control group. As this is an intervention study, thus blinding is not applicable for data collection personnel and participants. The health clinics that involved in this study will be maternal and child health clinics.

This study will use a set of questionnaires to obtain information on personal information, anthropometry data, prenatal knowledge, physical activity, psychosocial well-being, dietary intake, quality of life, sleep quality and gestational weight gain of the subjects, based on appropriate instruments. Re-assessment will be performed at month-6 and month-9 (delivery) after baseline measurements. During the re-assessment, the data will be collected again on dietary intake, physical activity, psychosocial well-being, sleep quality and quality of life. All subjects will be followed up prospectively until delivery. The follow up data collection will be matched with the prenatal visit of the pregnant mother to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian women
* 18 - 40 years old
* Single pregnancy
* At first trimester or second trimester
* All ethnicities
* Meet or did not meet with dietitian before
* With or without diseases (diabetes mellitus with/ without low dose insulin, hypertension, hyperlipidaemia, overweight/ obese)
* Own smart phone with internet access
* All BMI categories

Exclusion Criteria:

* Diagnosed by medical doctor with major psychiatric problems (bipolar depression, schizophrenia, suicidal risk)
* Multiple pregnancies
* On other intervention program
* Grand multipara
* Severe comorbidities (cardiac diseases, severe anaemia)
* Type 1 diabetes mellitus or Type 2 diabetes mellitus with high dose insulin

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 294 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Gestational Weight Gain | 3 points time (Baseline, 6th month, 9th month/ delivery)
  Weight gain (kg)

SECONDARY OUTCOMES:
Prenatal knowledge | 1 point1 time (Baseline)
  The maternal health literacy inventory in pregnancy (MHELIP)
  MHELIP score to 4 categories: 'inadequate', 'problematic' (which together also define 'limited' health literacy), 'sufficient and 'excellent' (which together also defined 'desired' health literacy):
  Inadequate= 0-50 Problematic= 50.1-66 Sufficient= 66.1-84 Excellent=84.1-100
Physical activity | 2 points time (Baseline, 6th month)
  Pregnancy Physical Activity Questionnaire (PPAQ)
  The activity was classified by intensity: sedentary (< 1.5 METs), light (1.5- < 3.0 METs), moderate (3.0-6.0 METs) or vigorous (> 6.0 METs) and the average number of MET-hours per week expended in each intensity level was calculated. The higher the score, the more active the subject is.
Psychosocial well-being | 3 points time (Baseline, 6th month, 9th month/ delivery)
  Depression Anxiety and Stress Scale (DASS-21)
  Scores on the DASS-21 will need to be multiplied by 2 to calculate the final score.
  Depression (Normal: 0-9; Mild: 10-13; Moderate: 14-20; Severe: 21-27; Extremely Severe: 28+) Anxiety (Normal: 0-7; Mild: 8-9; Moderate: 10-14; Severe: 15-19; Extremely Severe: 20+) Stress (Normal: 0-14; Mild: 15-18; Moderate: 19-25; Severe: 26-33; Extremely Severe: 34+)
Nutritional status | 3 points time (Baseline, 6th month, 9th month/ delivery)
  24-hour dietary recall (2 weekdays and 1 weekend)
Quality of life (well being) | 3 points time (Baseline, 6th month, 9th month/ delivery)
  WHO 5 item well being index
  The raw score is calculated by totalling the figures of the five answers. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
  To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life.
Sleep quality | 3 points time (Baseline, 6th month, 9th month/ delivery)
  Pittsburgh Sleep Quality Index (PSQI)
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Pregnancy outcome (Type of delivery) | 1 point time (9th month/ delivery)
  Spontaneous vaginal delivery (SVD): Cephalic/ Breech/ Assisted Breech; Instrumental Delivery: Forceps/ Vacuum; Caesarean: Elective/ Emergency/ Lower segment Caesarean section (LSCS)/ Classical
Pregnancy outcome (Apgar Score) | 1 point time (9th month/ delivery)
  @1 minute and @5 minutes (Apgar Score 7-10: Good outcome)
Pregnancy outcome (Born term) | 1 point time (9th month/ delivery)
  Yes / No (_______ week)
Pregnancy outcome (Infant weight) | 1 point time (9th month/ delivery)
  weight (kg)
Pregnancy outcome (Infant length) | 1 point time (9th month/ delivery)
  length (cm)
Pregnancy outcome (Infant head circumference) | 1 point time (9th month/ delivery)
  head circumference (cm)
Pregnancy outcome ( Infant breast circumference) | 1 point time (9th month/ delivery)
  breast circumference (cm)
Pregnancy outcome (Infant gender) | 1 point time (9th month/ delivery)
  Male/ Female
Pregnancy outcome (Maternal complications) | 1 point time (9th month/ delivery)
  Postpartum hemorrhage (PPH)/ Eklampsia / Retained placenta/ Venous thromboembolism (VTE)/ Postpartum depression
Pregnancy outcome (Infant complications) | 1 point time (9th month/ delivery)
  Miscarriage/ Prematurity/ Stillbirth/ Congenital anomalies/ Shoulder dystosia/ Jaundice / Respiratory related / Transient Tacypnoiec of newborn (TTN)/ Pneumonia (lung infection)

CONTACTS AND LOCATIONS:
Overall Officials: Yoke Mun Chan, Principal Investigator — Universiti Putra Malaysia
Locations (3):
- Malaysia (3):
  - Seri Kembangan Health Clinic, Seri Kembangan, Selangor
  - Presint 18 Health Clinic, Putrajaya
  - Presint 9 Health Clinic, Putrajaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Er YT, Chan YM, Mohd Shariff Z, Abdul Hamid H, Mat Daud Z', Yong HY. Dietitian-led cluster randomised controlled trial on the effectiveness of mHealth education on health outcomes among pregnant women: a protocol paper. BMJ Open. 2023 Nov 20;13(11):e075937. doi: 10.1136/bmjopen-2023-075937. PMID 37989361